CLINICAL TRIAL: NCT01818947
Title: A Multicentre, Retrospective Chart Review Study to Characterise Gefitinib Usage and Outcomes in Routine Treatment
Brief Title: Gefitinib Usage and Outcomes in Routine Treatment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OGB-IRE-2012/1
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; epidermal growth factor receptor mutation; gefitinib; Iressa
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gefitinib

SUMMARY:
The purpose of this study is to understand real world gefitinib usage patterns, patient characteristics and outcomes and to present these for a Caucasian population

DETAILED DESCRIPTION:
A multicentre, retrospective chart review study to characterise gefitinib usage and outcomes in routine treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients who received gefitinib first line in the UK Single Payment Access (SPA) scheme
* Locally advanced or metastatic EGFR mutation positive NSCLC
* Supplied with first pack of gefitinib prior to 1st January 2012

Exclusion Criteria:

* Patient was treated privately (i.e. outside the NHS)
* Gefitinib was second-line therapy following treatment failure on a prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital clinic
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Assessment of treatment duration, as a surrogate of Clinical Benefit (CB) in a 'Real World' population treated with gefitinib | 6 months
  Retrospective population [2009 to 2013]
Assessment of Overall Survival (OS) in a 'Real World' population treated with gefitinib | 6 months
  Retrospective population [2009 to 2013]

SECONDARY OUTCOMES:
Assessment of Overall Survival (OS) in the subgroup of patients of Caucasian ethnicity and in the subgroup of patients treated with gefitinib for at least 3 months | 6 months
  Retrospective population [2009 to 2013]
Assessment of Treatment duration in the subgroup of patients of Caucasian ethnicity and in the subgroup of patients treated with gefitinib for at least 3 months | 6 months
  Retrospective population [2009 to 2013]
Characteristics of patients treated with gefitinib for all patients and stratified by whether gefitinib discontinued treatment before or after three months | 6 months
  Retrospective population [2009 to 2013]
Description of treatment patterns in patients treated with gefitinib (prior chemo, treatment breaks, treatment on discontinuation) | 6 months
  Retrospective population [2009 to 2013]
Duration of treatment in patients stratified by age, gender, stage and performance status. | 6 months
  Retrospective population [2009 to 2013]
Overall Survival (OS) in patients stratified by age, gender, stage and performance status. | 6 months
  Retrospective population [2009 to 2013]

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Blackhall, MBCHB FRCP, Principal Investigator — The Christie NHS Foundation Trust
Locations (12):
- United Kingdom (12):
  - Queen Elizabeth Hospital, Birmingham
  - Velindre Nhs Trust, Cardiff
  - Harrogate District Hospital, Harrogate
  - Leeds Teaching Hospitals, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Mount Vernon Hospital Nhs Trust, London
  - Royal Marsden Hospital, London
  - University College Hospital, London
  - Christie Hospital Nhs Trust, Manchester
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Northern General Hospital, Sheffield
  - York District Hospital, York